CLINICAL TRIAL: NCT06784817
Title: Investigating the Periodontal Status of Traditional and Heated Tobacco Product Users: A Cross-sectional Observational Study
Brief Title: Investigating the Periodontal Status of Traditional and Heated Tobacco Product Users
Acronym: INPER-THT
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Collaborators: Center for Translational Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: SE RKEB 131/2023
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-09

CONDITIONS: Gingivitis and Periodontal Diseases
Keywords: smoking; heated tobacco products; periodontal diseases
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Gingival crevicular fluid samples will be collected from the deepest periodontal pocket on the buccal aspects of the mesial or distal interproximal sites of a maxillary single rooted tooth. A sterile paper strip (Periopaper, Amityville, NY, USA) is placed in the periodontal sulcus until resistance is felt and then held in place for 30 seconds. The strips of paper are then immediately placed in a calibrated electronic gingival fluid measuring device (Periotron 8000, Oraflow. Inc., New York) for volume determination (μL).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Non-smokers: Never consumed tobacco in any form
- Cigarette smokers: Smoking at least 1 cigarette daily for at least 12 months
- Heated tobacco product users: Using heated tobacco products e.g. IQOS exclusively at least once daily in the past 12 months and was not a regular traditional cigarette smoker

SUMMARY:
This cross-sectional observational study aims to compare the clinical and radiographic periodontal status, as well as gingival crevicular fluid volume, among cigarette smokers, heated-tobacco product users, and non-smokers. Specifically, the aim is to determine whether tobacco product users exhibit worse clinical parameters-such as probing pocket depth, bleeding on probing, plaque index, clinical attachment loss-along with greater radiographic bone loss and higher gingival crevicular fluid volume than non-smokers.

DETAILED DESCRIPTION:
Smoking is one of the main risk factors of periodontitis and its harmful effects on periodontal health are now well known. Thanks to worldwide restrictions, the use of traditional cigarettes is declining, but new alternative tobacco products such as heated tobacco products (e.g. IQOS, glo) have appeared on the market. These devices are often perceived less harmful by consumers, but there are conflicting results in the literature regarding their health effects.

Only one study has assessed periodontal health in heated tobacco product users, but in this study all participants were former smokers. No studies have evaluated periodontal health in heated tobacco users without a history of smoking traditional cigarettes on a regular basis.

Therefore, the aim of the present cross-sectional observational study is to compare the clinical and radiographic periodontal status and gingival crevicular fluid (GCF) volume among cigarette-smokers, heated-tobacco product users and non-smokers.

The null hypothesis is that different tobacco product users have worse clinical and radiological periodontal parameters and higher GCF volume than non-smokers.

The study will be performed at the Department of Prosthodontics at Semmelweis University, Budapest, Hungary. Patients will be enrolled from the patient material of the Department of Prosthodontics.

ELIGIBILITY:
Inclusion Criteria:

* Smokers who smoke at least one cigarette daily for the past 12 months.
* Exclusive users of heated tobacco products (e.g., IQOS), using them at least once daily for the past 12 months and not regular traditional cigarette smokers.
* Non-smokers who have never consumed tobacco in any form.

Exclusion Criteria:

* Users of electronic cigarettes, smokeless tobacco, waterpipes, or any other tobacco products.
* Dual users of tobacco products.
* Individuals diagnosed with systemic diseases.
* Edentulousness or severe tooth loss (fewer than 20 remaining teeth).
* Individuals who have taken antibiotics, steroids, or non-steroidal anti-inflammatory drugs in the past 90 days.
* Pregnant or breastfeeding women.
* History of periodontitis.
* Individuals refusing to sign the written informed consent form.
* Third molars are excluded from examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy induviduals with no systemic diseases will be selected for this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss in mm ( MBL) | At baseline (first visit)
  Digital periapical radiographs will be taken of each tooth and be viewed on a calibrated computer screen using a software program. MBL is defined as the vertical distance from 2 mm below the cemento-enamel junction (CEJ) to the most crestal part of marginal alveolar bone.
  Measures of effect: mean and standard deviation

SECONDARY OUTCOMES:
Full mouth plaque index (PI) | At baseline (first visit)
  It is measured at 6 sites per tooth (mesio-buccal, mid-buccal, disto-buccal,disto-lingual/palatal, mid-lingual/palatal and mesio-lingual/palatal) on all maxillary and mandibular teeth, except third molars. It is measured dichotomously. Score 1 if plaque biofilm is present and 0 if plaque biofilm is absent. A percentage score for the whole mouth is obtained by adding together the values for all teeth, dividing by the number of teeth and multiplying the result by 100.
  Measures of effect: mean and standard deviation
Bleeding on Probing (BOP) | At baseline (first visit)
  It is measured at 6 sites per tooth (mesio-buccal, mid-buccal, disto-buccal,disto-lingual/palatal, mid-lingual/palatal and mesio-lingual/palatal) on all maxillary and mandibular teeth, except third molars. It is measured dichotomously. Score 1 if bleeding is present and 0 if bleeding is absent. A percentage score for the whole mouth is obtained by adding together the values for all teeth, dividing by the number of teeth and multiplying the result by 100.
  Measures of effect: mean and standard deviation
Probing Pocket Depth (PPD) | At baseline (first visit)
  It is measured at 6 sites per tooth (mesio-buccal, mid-buccal, disto-buccal,disto-lingual/palatal, mid-lingual/palatal and mesio-lingual/palatal) on all maxillary and mandibular teeth, except third molars. Using an UNC-15 periodontal probe, the distance from the gingival margin to the base of the periodontal pocket or sulcus is measured. This is recorded in millimeters (mm). Measures of effect: mean and standard deviation
Clinical attachment level (CAL) | At baseline (first visit)
  It is measured at 6 sites per tooth (mesio-buccal, mid-buccal, disto-buccal,disto-lingual/palatal, mid-lingual/palatal and mesio-lingual/palatal) on all maxillary and mandibular teeth, except third molars. To calculate the CAL, the position of the gingival margin relative to the cementoenamel junction (CEJ) and the probing pocket depth is added together. CAL ismeasured in millimeter to the nearest mm using UNC-15 periodontal probe. Measures of effect: mean and standard deviation
Gingival Crevicular Fluid (GCF) volume in μL | At baseline (first visit)
  GCF samples are taken from the deepest periodontal pocket on the buccal aspects of the mesial or distal interproximal sites of a maxillary single rooted tooth. Prior to GCF collection, the selected site is isolated with sterile cotton swabs and the supragingival oral biofilm is carefully removed. The tooth is then dried with a gentle air. A sterile paper strip (Periopaper, Amityville, NY, USA) is placed in the periodontal sulcus until resistance is felt and then held in place for 30 seconds. Samples contaminated with blood or saliva are discarded and a new sample is taken from the same site after 15 minutes. The strips of paper are then immediately placed in a calibrated electronic gingival fluid measuring device (Periotron 8000, Oraflow. Inc., New York) for volume determination.
  Measures of effect: mean and standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Kispélyi, Dental, Study Director — Semmelweis University, Department of Prosthodontics; Kata Kelemen, Dental, Study Director — Semmelweis University, Department of Prosthodontics; Brigitta Teutsch, Medical doctor, Study Chair — Center for Translational Medicine, Semmelweis University
Locations (1):
- Semmelweis University Department of Prosthodontics, Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No
All data supporting our findings will be found in the prepared manuscript and the supplementary material.